CLINICAL TRIAL: NCT00774371
Title: The Survivors' Health And Physical Exercise Study
Brief Title: Weight Reduction Intervention for Breast Cancer Survivors
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Cancer Society, Inc. (Other); San Diego State University (Other)
Responsible Party: Principal Investigator, Cheryl Rock, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSGPB-04-258-01-CPPB; UCSD ID# 2004-2839
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Overweight; Obese; Breast cancer survivors; Weight loss; Physical activity; Exercise; Cognitive behavioral therapy
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity; Weight Loss; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Weight list control group was the comparison to the immediate treatment group.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The intervention program consists of group sessions provided according to the following schedule: weekly for 4 months, every other week for two months, and follow-up monthly sessions through 18 months of active subject participation. The time points for data collection from all subjects are baseline, 6 months, and 18 months. The group sessions offered to the treatment study arm are closed-group contingents with an average of 12-15 women assigned to each group.
  Interventions: Behavioral: Cognitive behavioral therapy CBT) for weight loss

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy CBT) for weight loss — The intervention program emphasizes regular physical activity, healthy eating, and psychological components within the structure of CBT for obesity. The physical activity component emphasizes planned aerobic exercise, increased physical activity and strength training. A deficit of 500-1000 kcal/day is the recommended level of dietary modification to promote weight loss and maintenance. Group sessions are held weekly for 4 months, every other week for two months, and monthly sessions through 18 months. Data are collected at baseline, 6 months, and 18 months. Wait-list group subjects will receive general contact without specific reference to weight management topics through a 24-month period of data collection and will then be provided intervention materials in a seminar format.

SUMMARY:
Overweight or obesity is an established negative prognostic factor in both premenopausal and postmenopausal breast cancer. Several mechanisms have been proposed to explain the adverse effect of excess body fat on prognosis following the diagnosis of breast cancer, including increased circulating sex hormones, insulin, leptin, and various growth factors. Results from previous studies suggest that specific strategies can facilitate weight reduction and maintenance of weight loss in this target population. This randomized clinical trial will recruit 253 overweight or obese women who have been previously treated for early stage breast cancer and will test whether a multifaceted approach to promoting healthy weight management can achieve the goal of weight loss and maintenance. Additionally, this study tests whether weight loss is associated with changes in biological and psychosocial factors, including eating attitudes and behaviors and health-related quality of life. The intervention incorporates cognitive-behavioral therapy, increased physical activity, diet modification to facilitate a modest reduction in energy intake, and strategies to improve body image and self-acceptance. This approach and intervention have been pilot-tested with breast cancer survivors in a developmental project, which resulted in the intervention group losing significantly more weight than the wait-list control group.

Study Aims include: testing whether an intervention that emphasizes increased physical activity and individualized diet modification to promote an energy imbalance is associated with a greater degree of weight loss and maintenance of that loss over an 18-month time period; describing the effect of the intervention on hormones and growth factors; describing the relationships between body weight and weight reduction and measures of selected psychosocial factors. Measurements of hormonal and psychosocial factors in this study will provide insight into the responsiveness of these factors to weight loss in overweight or obese breast cancer survivors, which will provide an indication of the degree of clinical benefit that is achieved with the intervention efforts. Results from this study may enable the development of broader efforts transferable to clinical practice and public health, and thus, may ultimately have a substantial effect on the risk for recurrence and long-term survival of the estimated 1.98 million breast cancer survivors in the U.S. today.

DETAILED DESCRIPTION:
Background: Overweight or obesity is an established negative prognostic factor in both premenopausal and postmenopausal breast cancer. Adverse effects of adiposity on prognosis may be explained by effects on gonadal hormones, insulin, insulin-like growth factor (IGF)-I, IGF binding proteins (IGFBPs), and leptin.

Objective/Hypothesis: This study tests whether a multifaceted approach can achieve weight loss and maintenance in overweight or obese breast cancer survivors. The intervention incorporates cognitive-behavioral therapy, increased physical activity, diet modification, and strategies to improve body image and self-acceptance. This approach and intervention were developed and pilot-tested with support from a previous peer-reviewed grant. Weight change from baseline to one year in the pilot study (n=85) was -5.2 (6.3) kg (mean [SD]) in the intervention group vs. -0.1 (6.5) kg in the control group (P < 0.05), using intent to treat analysis with baseline values carried forward for dropouts.

Specific aims: (1) To test whether the intervention promotes weight loss and maintenance of that loss over an 18-month time period in a larger group; (2) To describe the effect of the intervention on hormonal factors (insulin, leptin, IGF-I, IGFBP-1, IGFBP-3, sex-hormone binding globulin, and serum estrogens); and (3) To describe the relationships between body weight and weight reduction and measures of psychosocial factors (health-related quality of life, fatigue, depression, eating attitudes, and weight and shape concerns).

Study design: The study targets 253 overweight or obese women previously treated for early stage breast cancer and utilizes a randomized study design with subjects assigned to the group-based healthy weight management program (with individualized telephone counseling support) or a wait-list control group. Data collection includes anthropometric and psychosocial measures, body composition (dual-energy x-ray absorptiometry), cardiopulmonary fitness testing, and hormonal measures at baseline and six and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Stage I-IIIA breast cancer within the previous 10 years
* Have completed initial treatments (i.e., surgery, adjuvant chemotherapy, radiation therapy)
* Have initial BMI >25.0 kg/m2
* A minimum of 15 kg over ideal weight
* Willingness and ability to attend group meetings and to maintain contact with the investigators for 18 months
* Ability to provide dietary and exercise data by telephone at prescribed intervals.

Exclusion Criteria:

* Inability to participate in physical activity because of severe disability

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2005-01; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 2 years

SECONDARY OUTCOMES:
Increase in physical activity levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L. Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Rock CL, Pande C, Flatt SW, Ying C, Pakiz B, Parker BA, Williams K, Bardwell WA, Heath DD, Nichols JF. Favorable changes in serum estrogens and other biologic factors after weight loss in breast cancer survivors who are overweight or obese. Clin Breast Cancer. 2013 Jun;13(3):188-95. doi: 10.1016/j.clbc.2012.12.002. Epub 2013 Jan 29. PMID 23375717
- See also: Related Info — http://nutritionandweightcontrol.ucsd.edu/